CLINICAL TRIAL: NCT04970680
Title: Comparison Between Two Techniques of Percutaneous Peristyloid Glossopharyngeal Block as an Analgesic Tool After Tonsillectomy
Brief Title: Percutaneous Peristyloid Glossopharyngeal Block After Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: glossopharyngeal nerve block
Record Dates: First submitted 2021-03-08; First posted 2021-07-21 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Pain
Keywords: analgesia; tonsillectomy
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: two groups, each will have peristyloid glossopharyngeal block, one with the help of ultrasound technology and the other blindly
Who Masked: Participant, Outcomes Assessor
Masking Description: the participant will have the block while anaesthetized, the care provider will do the block either blindly or using ultrasonic, the outcome assessor will not know which one have which technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- blind glossopharyngeal nerve block (Active Comparator): patients will have the glossopharyngeal nerve block with the blind technique
  Interventions: Procedure: glossopharyngeal nerve block
- ultrasonic glossopharyngeal nerve block (Active Comparator): patients will have the glossopharyngeal nerve block using the ultrasonic technique
  Interventions: Procedure: glossopharyngeal nerve block

INTERVENTIONS:
Procedure: glossopharyngeal nerve block — glossopharyngeal nerve block either blindly or using the ultrasonic technique

SUMMARY:
Adenotonsillectomy surgery in paediatrics is commonly managed as an ambulatory surgery. This may be attributed to the use of the electro-dissection surgical technique that decreases the incidence of immediate postoperative haemorrhage. However, the use of the electro-cautery technique increases postoperative inflammation.

This study aimed to compare the glossopharyngeal nerve block using the blind technique with the use of the ultrasound guidance Primary: FLACC score in the two groups 0,2,4,6 h after surgery at rest and with swallowing Secondary: need to analgesics, the difficulty of the technique, time consumption, recovery time, surgeon satisfaction, parents satisfaction, staff nurse satisfaction, anaesthetist self-confidence

DETAILED DESCRIPTION:
INTRODUCTION Adenotonsillectomy surgery in paediatrics is commonly managed as an ambulatory surgery. This may be attributed to the use of the electro-dissection surgical technique that decreases the incidence of immediate postoperative haemorrhage. However, the use of the electro-cautery technique increases postoperative inflammation.

Sensory fibres of the glossopharyngeal nerve supply the tonsillar and peri-tonsillar areas. Thus, a bilateral glossopharyngeal nerve block may alleviate post-tonsillectomy pain and improve postoperative analgesia.

This is a Prospective randomized controlled clinical study, to compare two different technique used to block the glossopharyngeal nerve.

AIM OF WORK To improve post tonsillectomy pain control in children Anaesthesia, postoperative analgesia Paediatrics 3-7 years Tonsillectomy NOT adenotonsillectomy Postoperative control of pain OBJECTIVES This study aimed to compare the glossopharyngeal nerve block using the blind technique with the use of the ultrasound guidance Primary: FLACC score in the two groups 0,2,4,6 h after surgery at rest and with swallowing Secondary: need to analgesics, the difficulty of the technique, time consumption, recovery time, surgeon satisfaction, parents satisfaction, staff nurse satisfaction, anaesthetist self-confidence METHODOLOGY 54 ASA I children allocated randomly into two groups: Group BL: Blind percutaneous peristyloid injection Group US: ultrasound-guided percutaneous peristyloid glossopharyngeal nerve block 54 children aged 3 to 7 years undergoing adenotonsillectomy without adenoidectomy were randomized to receive either local blind percutaneous peistyloid glossopharyngeal nerve block (n=27) or the use of ultrasound guidance for the same block (n=27). The pain was assessed by the FLACC scale or Face, Legs, Activity, Cry, Consolability scale, need for analgesics, and acceptance of diet during the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* children aged 3-7 years
* scheduled for tonsillectomy

Exclusion Criteria:

* younger or elder children
* associated adenoidectomy
* history of allergy to local anaesthetics

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
change in face, legs, activity, cry, and consolability (FLACC) score | Immediately postoperatively considered as 0 hour, then at 2 hours, again at 4 hours, and lastly at 6 hours after surgery all measures will be both at rest and with swallowing
  FLACC is a behavioural pain assessment scale used for nonverbal or preverbal patients who cannot self-report their pain level. Pain is assessed through observation of 5 categories including the face, legs, activity, cry, and consolability. The scale ranges from 0 to 10 where 0 records for no pain and 10 records for the worst pain

SECONDARY OUTCOMES:
need for postoperative analgesia | immediately postoperatively considered as 0 hour, then at 2 hours, again at 4 hours, and lastly at 6 hours after surgery
  need to analgesics in doses and frequencies both at rest and with swallowing.
difficulty of the technique | immediately after the intervention
  prescribed by the operator either easy or difficult
time consumption | immediately after the intervention
  from the start of preparation of the procedure, till the end of the block time in minutes
recovery time | immediately before shifting the patient to recovery room
  from the end of the surgery, till shifting the patient from operation table to recovery bed time in minutes
surgeon satisfaction assessed by visual analogue scale (VAS) | immediately after discharging the patient to home
  described by the surgeon him self on a scale ranging from very satisfactory to unsatisfactory
anesthetists self-confidence | immediately after the intervention
  described as yes or no
parents satisfaction | immediately before discharging the patient to home
  described by the parents on a scale ranging from very satisfactory to unsatisfactory
staff nurse satisfaction | immediately before shifting the patient from the recovery room to the day care unite by recovery nurse, and immediately after discharging the patient to home by daycare unite nurse
  described by the recovery nurse and daycare unite nurse on a scale ranging from very satisfactory to unsatisfactory

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided